CLINICAL TRIAL: NCT00323232
Title: Two-Hole Versus Four-Hole Dynamic Hip Screw (DHS) for the Treatment of Intertrochanteric Fractures: A Prospective Randomized Trial
Brief Title: Comparison of Treatment Outcomes in Hip Fractures Surgically Fixed With Either a Two or Four Hole Device.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Dr. P J O'Brien, University of British Columbia
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C05-0441
Record Dates: First submitted 2006-05-08; First posted 2006-05-09 (Estimated); Last update posted 2011-04-27 (Estimated); Status verified 2011-04

CONDITIONS: Hip Fracture
Keywords: DHS, Intertrochanteric
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: 2 Versus 4 Hole DHS — See Detailed Description.

SUMMARY:
Although Standard of Care for Hip Fractures is the Device (Dynamic Hip Screw) being studied in this project, and both sizes (the 2 and the 4 hole versions) are currently in use there is not widespread agreement yet whether there is an optimal number of screws (2 or 4) required for the best outcomes. If it can be shown that a 2 hole version is just as successful in outcomes it would allow for a smaller incision (surgical cut) at the site of the fracture. This could reduce soft tissue dissection, operating time, and surgical blood loss. This in turn would reduce post operative pain, blood loss, and hospital length of stay.

DETAILED DESCRIPTION:
This study has been designed to prospectively evaluate the clinical results of a two-hole versus four-hole dynamic hip screw in the treatment of intertrochanteric fractures.

It is estimated that over 27,000 hip fractures occur in Canada each year, at an estimated cost of $10,000 per patient per hospitalization. Intertrochanteric hip fractures account for approximately half of all hip fractures. While many surgical treatment options exist, the accepted standard fixation device for the treatment of both stable and unstable intertrochanteric hip fractures is the dynamic hip screw.

No consensus exists regarding the optimal number of screws required for adequate side plate fixation for the treatment of intertrochanteric fractures. The most commonly used device is the 135-degree four-hole side plate, however, decreasing the length of the side plate would theoretically allow for a smaller incision site, minimal soft-tissue dissection, shortened operating time, and reduced operative blood loss. This in turn would reduce post-operative pain, blood loss, and length of hospital stay. With the majority of hip fractures occurring in the frail, elderly population, a less invasive procedure potentially decreases overall patient mortality.

Biomechanical studies simulating stable and unstable intertrochanteric fractures have suggested that fewer screws are adequate for good side plate fixation. Two clinical trials have reviewed series of fractures treated with a two-hole DHS and have reported favorable results. No prospective randomized study to date, however, has directly compared the clinical results of the standard four-hole plate with that of the two-hole plate. We propose a study is to evaluate the clinical results of the two-hole versus four-hole plate for the treatment of intertrochanteric fractures with a minimum 6-month follow-up.

This study's aim is to develop clinical outcome data which can be used (a) determine range of expected clinical outcomes resulting from current standard management of these injuries, and (b) as the basis of reporting on the clinical outcomes of these injuries in the peer-reviewed literature.

Patients over the age of 65 who have sustained an isolated 2-, 3-, and 4-part intertrochanteric hip fractures will be included in this study.

Patients who have Pathological, subtrochanteric, reverse obliquity fractures, multiple injuries, and patients whose time to the operating room exceeds 48 hours will be excluded.

The primary outcome measure to be assessed is mechanical failure of fixation. Secondary variables to be assessed during the hospital stay are: length of incision, post-operative pain, analgesic use, operative time, and mean hemoglobin drop. Length of hospital stay and medical complications will also be assessed.

They will subsequently be followed at six weeks, 3 months, and six months post-operatively in clinic with a physical exam and a pelvis and hip radiograph, and an inquiry will be made as to their general medical condition and any significant medical complications since discharge. A functional inquiry and quality of life score will be administered pre-operatively and at each subsequent clinic visit.

ELIGIBILITY:
Inclusion Criteria:

Consenting patients over the age of 65 with an isolated 2-, 3-, and 4-part intertrochanteric hip fractures will be included in this study.

Exclusion Criteria:

-

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Mechanical failure of fixation (up to 6 months)

SECONDARY OUTCOMES:
Length of incision, post-operative pain, analgesic use, operative time, and mean hemoglobin drop. Length of hospital stay and medical complications will also be assessed while hospitalized

CONTACTS AND LOCATIONS:
Overall Officials: P J O'Brien, MD, Principal Investigator — The University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada